CLINICAL TRIAL: NCT00851435
Title: A Non-comparative Open Pilot Trial to Assess the Safety and Pharmacokinetics of up to Three Single Doses of AERUMAB 11 (KBPA-101) in Patients With Hospital Acquired Pneumonia Caused by Serotype O11 P. Aeruginosa
Brief Title: Safety and Pharmacokinetics of KBPA-101 in Hospital Acquired Pneumonia Caused by O11 Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kenta Biotech Ltd (Industry)
Responsible Party: Violetta Georgescu, Kenta Biotech Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-101-002
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pneumonia; Ventilator Associated Pneumonia
Keywords: Pneumonia; Nosocomial pneumonia; Pseudomonas aeruginosa; Monoclonal antibody; Hospital-Acquired Pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Pseudomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KBPA-101, a monoclonal antibody (Experimental): 1.2 mg/kg KBPA-101 i.v. infusion, 3 single doses, every third day
  Interventions: Biological: KBPA-101

INTERVENTIONS:
Biological: KBPA-101 — 1.2 mg/kg KBPA-101 i.v. infusion, 3 single doses, every third day

SUMMARY:
The objectives of this open study are to assess the safety, tolerability, pharmacokinetics and clinical outcome of patients who have HAP caused by Pseudomonas aeruginosa serotype O11 after three separate administrations of KBPA-101 every third day in addition of standard of care antibiotic treatment.

DETAILED DESCRIPTION:
Hospital acquired pneumonia (HAP) is a pneumonia occurring 48 hours or more after hospital admission. HAP occurs in patients on conventional hospital wards and in intensive care units (ICU), some of them associated to mechanical ventilation, known as Ventilator Associated Pneumonia (VAP). VAP is the most common infection on intensive care units representing 82% of HAP cases. Pseudomonas aeruginosa is one of the most frequent pathogens involved in ICU-HAP and despite of adequate treatment its crude mortality remains as high as 70% of the cases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Patients under intensive care management with hospital acquired pneumonia
* Microbiological diagnosis of P. aeruginosa serotype O11 HAP by lower respiratory tract specimen (BAL or miniBAL) and presence of a new or progressing pulmonary infiltrate, plus one of the three following criteria: a) fever greater than 38ºC, b) WBC greater than 10,000/mm3, or c) purulent sputum
* In non-intubated patients confirmed microbiological diagnosis of P. aeruginosa serotype O11 HAP by endotracheal aspirate (ETA) and modified clinical pulmonary infection score (CPIS) higher than 6 points
* Patient is expected to survive longer than 72 hours
* Written informed consent provided by the patient or by the relatives or the designated trusted person

Exclusion Criteria:

* Use of any investigational drug within 30 days preceding the first dose of KBPA-101, or planned use during the study and safety follow-up periods
* Existence of any surgical or medical condition that might render the patient unduly susceptible to possible toxicity from the monoclonal antibody, including septic shock with unstable hemodynamics,
* Patients with a known complement deficiency associated with systemic lupus erythematosus, paroxysmal nocturnal hemoglobinuria, hereditary angioedema, membranoproliferative glomerulonephritis, collagen vascular disease, autoimmune hepatitis, primary biliary cirrhosis, scleroderma, or recurrent Neisserial infections
* Confirmed Human Immunodeficiency Virus (HIV) infection
* Transplant patients and/or simultaneous treatment with systemic immuno-suppressive drugs.
* Patients with a known liver function deficiency, e.g. associated with liver cirrhosis (Child Pugh B or C) or acute hepatitis
* Administration of poly- or mono-immunoglobulins within the three months preceding the first dose of study drug or planned administration during the study period
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assessment of physical examination, laboratory parameters, vital signs, ECG and any adverse at repeated times since the screening phase till the end of the study. | 30 days

SECONDARY OUTCOMES:
To confirm the therapeutic plasma concentration of KBPA-101 | 30 days
To ascertain the therapeutic efficacy of KBPA-101 given in addition to standard care for hospital acquired pneumonia | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Violetta Georgescu, Study Director — Kenta Biotech Ltd
Locations (1):
- Several sites in Switzerland, France, Belgium and Greece, Basel, Switzerland